CLINICAL TRIAL: NCT00852020
Title: Safety, Tolerance and Efficacy of an Oral Nutritional Supplement in CHF and COPD Patients. A Randomised, Double-blind and Controlled Pilot Study.
Brief Title: Safety, Tolerance and Efficacy of an Oral Nutritional Supplement in Chronic Heart Failure and Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PCSU-002-CFS
Record Dates: First submitted 2009-02-13; First posted 2009-02-26 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cachexia; Chronic Obstructive Pulmonary Disease; Chronic Heart Failure
MeSH Terms: conditions — Cachexia; Pulmonary Disease, Chronic Obstructive | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): oral nutritional supplement containing n-3-fatty acids, amino acids and antioxidants
  Interventions: Dietary Supplement: oral nutrition supplement, food for special medical purposes
- 2 (Placebo Comparator): oral nutritional supplement (isocaloric, isonitrogenous)
  Interventions: Dietary Supplement: oral nutrition supplement, food for special medical purposes

INTERVENTIONS:
Dietary Supplement: oral nutrition supplement, food for special medical purposes — 2 servings of 200-300 ml per day, treatment period: 16 weeks

SUMMARY:
To test the compliance, tolerance, safety and to get preliminary insights into the efficacy of a new oral nutritional supplement (containing n-3 fatty acids, amino acids and antioxidants) designed to prevent or delay cachexia and anorexia in patients with chronic heart failure (CHF) or chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CHF or COPD
* current body weight less than 6 months ago
* BMI >=20 and <=30 kg/m2
* CHF: LVEF >=45% measured within the past 6 months
* symptom status equivalent to NYHA class II to IV
* biochemical abnormalities for total cholesterol, serum uric acid, abnormal high CRP
* on standard therapy of CHF including ACE inhibitors and beta blockers
* COPD: symptom status equivalent to GOLD standard class II to IV
* FEV1 < 80%
* FEV1/FEV < 70%

Exclusion Criteria:

* significant oedema in the time of screening and randomisation
* concomitant inflammatory diseases
* active infections including HIV and AIDS
* liver failure
* chronic renal failure (sCr>1.5mg/dL) or cardiac pacemaker
* acute or chronic infections
* insulin treated diabetes mellitus
* patient with established diagnosis of cachexia
* life expectancy of less than 6 months in the opinion of the investigator
* medications that impair sex hormone synthesis, secretion or function
* patients with psychiatric diseases
* body weight loss > 5% during the last 6 months or > 10% during the last 10 months
* suspected allergy to any component of the investigational product(s)
* fish oil supplementation within 3 months prior to the study entry
* taking vitamin supplements in doses greater than the Recommended Daily Allowances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
compliance to nutrition therapy | baseline, months 1, 2, 3, 4

SECONDARY OUTCOMES:
anorexia questionnaire | baseline, months 1, 2, 3, 4
Gastrointestinal syndrome score (GIS) | baseline, months 1, 2, 3, 4
body cell mass | baseline, months 1, 2, 3, 4
weight change | baseline, months 1, 2, 3, 4
hand grip strength | baseline, months 1, 2, 3, 4
patient global assessment (PGA) | baseline, months 2, 4

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Anker, Prof. MD PHD, Principal Investigator — Center of Cachexia Research, Department of Cardiology, Charité Campus Virchow-Klinikum, Berlin
Locations (4):
- Germany (2):
  - Center of Cachexia Research, Department of Cardiology, Charité, Campus Virchow-Klinikum, Berlin
  - Praxis für Pneumologie, Schwedt/Oder, Schwedt
- Poland (2):
  - Regionalne Centrum Leczenia Chorób Płuc i Alergii, NZOZ ALLMED, Piekary Śląskie
  - Specjalista Chorób Wewnętrznych Kardiolog, Ruda Śląska